CLINICAL TRIAL: NCT00335660
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Trial to Investigate the Safety and Efficacy of AV608 in Subjects With Idiopathic Detrusor Overactivity
Brief Title: Safety and Efficacy of AV608 in Subjects With Idiopathic Detrusor Overactivity
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Animal Safety Data
Sponsor: Avera Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AV608-106
Record Dates: First submitted 2006-06-08; First posted 2006-06-12 (Estimated); Last update posted 2008-02-25 (Estimated); Status verified 2008-02

CONDITIONS: Overactive Bladder Syndrome
Keywords: Idiopathic Detrusor Overactivity; NK-1 Receptor Antagonist; Neurokinin; Urge Incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge

INTERVENTIONS:
Drug: AV608

SUMMARY:
The purpose of this study is to assess the effects of AV608, a neurokinin 1 (NK-1) antagonist, in subjects with Idiopathic Detrusor Overactivity.

DETAILED DESCRIPTION:
This is a Phase 2, randomized, double-blind, placebo-controlled trial to evaluate the safety and efficacy of AV608 in subjects with idiopathic detrusor overactivity. Female subjects between 18 and 65 years of age with a diagnosis of Overactive Bladder Syndrome and urodynamic observation of involuntary detrusor contractions during the filling phase will be eligible for the trial.

Eligible subjects will complete a baseline urodynamic assessment. All subjects who participate in the study will receive 3 weeks of treatment with AV608 or placebo. At the end of the treatment period, subjects will complete a second urodynamic assessment.

ELIGIBILITY:
Inclusion Criteria:

* Female, 18 to 65 years of age, inclusive
* A current primary diagnosis of OAB
* Idiopathic detrusor overactivity, demonstrated by a urodynamic observation
* Evidence of frequency in combination with urinary urgency
* Written informed consent form
* Willingness to avoid pregnancy and practice adequate birth control
* Negative serum pregnancy test
* Agrees to refrain from blood donation during the course of the study

Exclusion Criteria:

* Subjects who are pregnant or lactating
* Clinically significant abnormality or clinically significant unstable medical condition
* QTc interval of 470 msec or greater at Visit 1
* Predominant stress urinary incontinence versus urge urinary incontinence based on subject history
* Neurogenic bladder (e.g. associated with spinal cord injury, multiple sclerosis, etc.)
* Anatomic or structural abnormalities possibly causing urinary incontinence or urgency, including but not limited to urogenital prolapse stage 2 or more according to the Pelvic Organ Prolapse Quantification (POP-Q) system
* Urological or gynecological surgery within 3 months of the baseline urodynamic assessment
* Current UTI or frequent UTIs (i.e., greater than or equal to 4 UTIs per year), interstitial cystitis, hematuria of unknown cause, or use of indwelling catheter
* Electro-stimulation therapy, bladder training, or physiotherapy for bladder control within 2 weeks of Visit 1
* History (within 1 year of Screening) of alcohol or substance dependence (except nicotine dependence) according to DSM-IV-TR criteria
* History of any kind of cancer within the last 2 years
* Existing non-malignant tumors that could compromise the function and/or anatomy of the lower urinary tract

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2006-06; Primary Completion 2007-06 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Comparison between treatment groups of the change from baseline in maximum cystometric bladder capacity

SECONDARY OUTCOMES:
Delay of the first involuntary detrusor contraction associated with symptomatic urgency
Urgency, frequency and urge incontinence events as recorded in the Subject Micturition Diary
Urgency Perception Scale

CONTACTS AND LOCATIONS:
Overall Officials: Linda Cardozo, MD FRCOG, Principal Investigator — King's College Hospital NHS Trust; Joao Siffert, MD, Study Director — Avera Pharmaceuticals, Inc.
Locations (13):
- Netherlands (3):
  - Amsterdam
  - Nieuwegein
  - Zeist
- United Kingdom (10):
  - Birmingham, England
  - Blackburn, England
  - Chertsey, England
  - Hull, England
  - Leeds, England
  - Liverpool, England
  - London, England
  - Plymouth, England
  - Sheffield, England
  - Falkirk, Scotland